CLINICAL TRIAL: NCT01608451
Title: Randomized Controlled Trial of Neo-adjuvant Progesterone and Vitamin D3 in Women With Large Operable Breast Cancer and Locally Advanced Breast Cancer.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual implies that clinical questions being questioned have lost its significance.
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Principal Investigator, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D3/377/TMH; TMH project No. 377 (Other: Tata Memorial Hospital)
Record Dates: First submitted 2012-05-22; First posted 2012-05-31 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Locally Advanced Breast Cancer and Large Operable Breast Cancer
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No additional treatment (No Intervention): No Injection Vit D3 or Injection Progesterone prior to chemotherapy cycle
- Inj. Proluton (Active Comparator): Injection Progesterone 500 mg deep IM before each cycle of NACT (for total 4 cycles) and one injection before surgery.
  Interventions: Drug: Inj. Progesterone
- Inj. Arachitol (Active Comparator): Injection Arachitol (Vitamin D3) 300,000 I.U/ml IM before each cycle of NACT (for total 4 cycles) and one injection before surgery.
  Interventions: Drug: Cholecalciferol
- Inj. Proluton and Inj. Arachitol (Active Comparator): Injection Arachitol (Vitamin D3) 300,000 I.U/ml IM and Injection Progesterone 500 mg deep IM before each cycle of NACT (for total 4 cycles) and one injection before surgery.
  Interventions: Drug: Cholecalciferol; Drug: Inj. Progesterone

INTERVENTIONS:
Drug: Cholecalciferol — Inj Arachitol 300,000 I.U/ml IM before each cycle of NACT (for total 4 cycles) and one injection before surgery.
  Other Names: IArachitol
  Arms: Inj. Arachitol; Inj. Proluton and Inj. Arachitol
Drug: Inj. Progesterone — Injection Progesterone 500 mg deep IM before each cycle of NACT (for total 4 cycles) and one injection before surgery.
  Other Names: Inj. Proluton Depot
  Arms: Inj. Proluton; Inj. Proluton and Inj. Arachitol

SUMMARY:
Randomized Controlled Trial of Neoadjuvant Progesterone and Vitamin D3 in women with Large Operable Breast Cancer and Locally Advanced Breast Cancer - A Feasibility Study

Primary Progesterone Timing of surgery during the menstrual cycle and its impact on survival in premenopausal women with operable breast cancer has been extensively researched and reinvestigated by Badwe et al in the randomized clinical trial of 'Primary Progesterone Therapy for Operable Breast Cancer' at Tata Memorial Hospital. The underlying assumption was that the presence of unopposed estrogen (in follicular phase) at the time surgery may be deleterious for survival and that circulating progesterone might counteract this deleterious effect.

Vitamin D3 The most prominent physiological role of hormonally active form of vitamin D3, 1,25-dihydroxyvitamin D3 (1,25(OH)2D3 or calcitriol), is regulation of calcium and phosphorous homeostasis and bone metabolism via an intracellular receptor (VDR) which is a member of steroid thyroid hormone super-family of receptors. The VDR receptors are also found in other tissues like breast and prostate.

Vitamin D compounds have also been implicated in promotion of apoptosis in breast cancer cells and evidence suggests that 1,25(OH)2D3 and its synthetic analogues may potentiate responsiveness of breast cancer cells to conventional cytotoxic agents.

Objectives

1. To see the effect of primary progesterone on survival in women with high risk breast cancer (large operable and locally advanced breast cancer)
2. To see the effect of Vitamin D3 as an antiproliferative, cytotoxic and apoptotic agent (negative growth regulator) by evaluation of surrogate markers of proliferation and apoptosis.

Inclusion Criteria:

* Unilateral breast cancer
* Large operable breast cancer/LOBC (T3N0M0 or T3N1M0) and Locally advanced breast cancer/LABC (T3N1-2M0; T2N2M0)
* Age <70 years
* Fit for CT

Exclusion Criteria:

* Prior Incision Biopsy or Excision Biopsy
* Metastatic breast cancer
* Renal failure or deranged Renal Function Test
* Hypoparathyroidism
* Pregnant or lactating mothers or women of childbearing age not practicing contraception
* Patient on any of the following drugs: Magnesium-containing antacids, Digitalis, Phenytoin barbiturates, Thiazide diuretics.
* Previous history of other cancers except cured skin and cervical carcinoma in situ.

Methodology / Treatment plan

The study drugs (Injectable Progesterone and Vitamin D3) will be tested in the neoadjuvant setting prior to administration of each chemotherapy cycle, in a 2x2 factorial design as below:

Neoadjuvant D3 will be administered as Inj. Arachitol 300,000 IU/ml intramuscular, before each chemotherapy cycle.

Neoadjuvant Progesterone used will be administered as single IM depot injection 500mg 5 days prior to each CT cycle and surgery date.

Primary Objectives Disease-free survival

Secondary Objectives Improvements in overall survival Tumor response

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer
* Large operable breast cancer/LOBC (T3N0M0 or T3N1M0) and Locally advanced breast cancer/LABC (T3N1-2M0; T2N2M0)
* Age <70 years
* Fit for CT

Exclusion Criteria:

* Prior IB or EB
* Metastatic breast cancer
* Renal failure or deranged RFT
* Hypoparathyroidism
* Pregnant or lactating mothers or women of childbearing age not practicing contraception
* Patient on any of the following drugs: Magnesium-containing antacids, Digitalis, Phenytoin barbiturates, Thiazide diuretics.
* Previous history of other cancers except cured skin and cervical carcinoma in situ.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival

SECONDARY OUTCOMES:
Improvements in overall survival, Tumor response | 5 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, MS (Surgery), Principal Investigator — Tata Memorial Hospital, Ernest Borges Road, Parel, Mumbai 400 012
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Hrushesky WJ, Bluming AZ, Gruber SA, Sothern RB. Menstrual influence on surgical cure of breast cancer. Lancet. 1989 Oct 21;2(8669):949-52. doi: 10.1016/s0140-6736(89)90956-2. PMID 2571865
- [Background] Badwe RA, Gregory WM, Chaudary MA, Richards MA, Bentley AE, Rubens RD, Fentiman IS. Timing of surgery during menstrual cycle and survival of premenopausal women with operable breast cancer. Lancet. 1991 May 25;337(8752):1261-4. doi: 10.1016/0140-6736(91)92927-t. PMID 1674070
- [Background] Heer K, Kumar H, Speirs V, Greenman J, Drew PJ, Fox JN, Carleton PJ, Monson JR, Kerin MJ. Vascular endothelial growth factor in premenopausal women--indicator of the best time for breast cancer surgery? Br J Cancer. 1998 Nov;78(9):1203-7. doi: 10.1038/bjc.1998.655. PMID 9820181
- [Background] Senie RT, Rosen PP, Rhodes P, Lesser ML. Timing of breast cancer excision during the menstrual cycle influences duration of disease-free survival. Ann Intern Med. 1991 Sep 1;115(5):337-42. doi: 10.7326/0003-4819-115-5-337. PMID 1863022
- [Background] Mathiasen IS, Colston KW, Binderup L. EB 1089, a novel vitamin D analogue, has strong antiproliferative and differentiation inducing effects on cancer cells. J Steroid Biochem Mol Biol. 1993 Sep;46(3):365-71. doi: 10.1016/0960-0760(93)90226-m. PMID 9831485
- [Background] Welsh J. Vitamin D and breast cancer: insights from animal models. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1721S-4S. doi: 10.1093/ajcn/80.6.1721S. PMID 15585794
- [Background] Gulliford T, English J, Colston KW, Menday P, Moller S, Coombes RC. A phase I study of the vitamin D analogue EB 1089 in patients with advanced breast and colorectal cancer. Br J Cancer. 1998 Jul;78(1):6-13. doi: 10.1038/bjc.1998.434. PMID 9662243
- [Background] Wang Q, Lee D, Sysounthone V, Chandraratna RAS, Christakos S, Korah R, Wieder R. 1,25-dihydroxyvitamin D3 and retonic acid analogues induce differentiation in breast cancer cells with function- and cell-specific additive effects. Breast Cancer Res Treat. 2001 May;67(2):157-68. doi: 10.1023/a:1010643323268. PMID 11519864
- [Background] Narvaez CJ, Zinser G, Welsh J. Functions of 1alpha,25-dihydroxyvitamin D(3) in mammary gland: from normal development to breast cancer. Steroids. 2001 Mar-May;66(3-5):301-8. doi: 10.1016/s0039-128x(00)00202-6. PMID 11179738
- [Background] James SY, Mackay AG, Colston KW. Effects of 1,25 dihydroxyvitamin D3 and its analogues on induction of apoptosis in breast cancer cells. J Steroid Biochem Mol Biol. 1996 Jul;58(4):395-401. doi: 10.1016/0960-0760(96)00048-9. PMID 8903423
- [Background] Vink-van Wijngaarden T, Pols HA, Buurman CJ, van den Bemd GJ, Dorssers LC, Birkenhager JC, van Leeuwen JP. Inhibition of breast cancer cell growth by combined treatment with vitamin D3 analogues and tamoxifen. Cancer Res. 1994 Nov 1;54(21):5711-7. PMID 7923220
- [Background] Sundaram S, Gewirtz DA. The vitamin D3 analog EB 1089 enhances the response of human breast tumor cells to radiation. Radiat Res. 1999 Nov;152(5):479-86. PMID 10521924
- [Background] Chaudhry M, Sundaram S, Gennings C, Carter H, Gewirtz DA. The vitamin D3 analog, ILX-23-7553, enhances the response to adriamycin and irradiation in MCF-7 breast tumor cells. Cancer Chemother Pharmacol. 2001 May;47(5):429-36. doi: 10.1007/s002800000251. PMID 11391859
- [Background] Sundaram S, Sea A, Feldman S, Strawbridge R, Hoopes PJ, Demidenko E, Binderup L, Gewirtz DA. The combination of a potent vitamin D3 analog, EB 1089, with ionizing radiation reduces tumor growth and induces apoptosis of MCF-7 breast tumor xenografts in nude mice. Clin Cancer Res. 2003 Jun;9(6):2350-6. PMID 12796405
- [Background] Zinser GM, Tribble E, Valrance M, Urben CM, Knutson JC, Mazess RB, Strugnell SA, Welsh J. 1,24(S)-dihydroxyvitamin D2, an endogenous vitamin D2 metabolite, inhibits growth of breast cancer cells and tumors. Anticancer Res. 2005 Jan-Feb;25(1A):235-41. PMID 15816543
- [Background] Muindi JR, Peng Y, Potter DM, Hershberger PA, Tauch JS, Capozzoli MJ, Egorin MJ, Johnson CS, Trump DL. Pharmacokinetics of high-dose oral calcitriol: results from a phase 1 trial of calcitriol and paclitaxel. Clin Pharmacol Ther. 2002 Dec;72(6):648-59. doi: 10.1067/mcp.2002.129305. PMID 12496746
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Cooper LS, Gillett CE, Patel NK, Barnes DM, Fentiman IS. Survival of premenopausal breast carcinoma patients in relation to menstrual cycle timing of surgery and estrogen receptor/progesterone receptor status of the primary tumor. Cancer. 1999 Nov 15;86(10):2053-8. doi: 10.1002/(sici)1097-0142(19991115)86:103.0.co;2-h. PMID 10570431
- [Background] Cooper LS, Gillett CE, Smith P, Fentiman IS, Barnes DM. Cell proliferation measured by MIB1 and timing of surgery for breast cancer. Br J Cancer. 1998 May;77(9):1502-7. doi: 10.1038/bjc.1998.247. PMID 9652769
- [Background] Saad Z, Bramwell VH, Wilson SM, O'Malley FP, Jeacock J, Chambers AF. Expression of genes that contribute to proliferative and metastatic ability in breast cancer resected during various menstrual phases. Lancet. 1998 Apr 18;351(9110):1170-3. doi: 10.1016/S0140-6736(97)07498-9. PMID 9643688
- [Background] Ferrieres G, Cuny M, Simony-Lafontaine J, Jacquemier J, Rouleau C, Guilleux F, Grenier J, Rouanet P, Pujol H, Jeanteur P, Escot C. Variation of bcl-2 expression in breast ducts and lobules in relation to plasma progesterone levels: overexpression and absence of variation in fibroadenomas. J Pathol. 1997 Oct;183(2):204-11. doi: 10.1002/(SICI)1096-9896(199710)183:23.0.CO;2-M. PMID 9390034
- [Background] Yang Q, Sakurai T, Yoshimura G, Suzuma T, Umemura T, Nakamura M, Nakamura Y, Mori I, Kakudo K. Prognostic value of Bcl-2 in invasive breast cancer receiving chemotherapy and endocrine therapy. Oncol Rep. 2003 Jan-Feb;10(1):121-5. PMID 12469156
- [Background] Harris AL, Zhang H, Moghaddam A, Fox S, Scott P, Pattison A, Gatter K, Stratford I, Bicknell R. Breast cancer angiogenesis--new approaches to therapy via antiangiogenesis, hypoxic activated drugs, and vascular targeting. Breast Cancer Res Treat. 1996;38(1):97-108. doi: 10.1007/BF01803788. PMID 8825127
- [Background] Viens P, Jacquemier J, Bardou VJ, Bertucci F, Penault-Llorca F, Puig B, Gravis G, Oziel-Taieb S, Resbeut M, Houvenaeghel G, Camerlo J, Birbaum D, Hassoun J, Maraninchi D. Association of angiogenesis and poor prognosis in node-positive patients receiving anthracycline-based adjuvant chemotherapy. Breast Cancer Res Treat. 1999 Apr;54(3):205-12. doi: 10.1023/a:1006112927565. PMID 10445419